CLINICAL TRIAL: NCT02785510
Title: Determining Clinical Profile of Parkinson's Disease Among Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Negida, (1) Principal Investigator; (2) Head of Scientific Committee, Student Research Unit, Zagazig University; and (3) Head of Scientific Committee, Egyptian National Research Collaborative., Zagazig University
Other Study IDs: Egy Neuro 1 study
Record Dates: First submitted 2016-05-22; First posted 2016-05-27 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Parkinson's disease is the second most common neurodegenerative disease affecting about 1-3% of population above 60 years. Recently, non-motor symptoms are getting more attention in PD management. The pattern of PD onset and clinical course differ from one population to another. Many studies have been conducted to determine the clinical profile of PD in populations worldwide. However, no similar studies have been conducted in Egypt. Therefore, the investigators will conduct a nation-wide, collaborative, cross sectional study to determine the pattern of Parkinson's disease onset, clinical course, and non-motor symptoms among Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the Parkinson's disease criteria of United Kingdom Brain Bank within the study centres.

Exclusion Criteria:

* Patients with vascular Parkinsonism (history of stroke)
* Patients with treatment induced Parkinsonism
* Patients with history of dopaminergic neurotoxin (1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet the diagnosis of Parkinson's disease according to the Parkinson's disease criteria of United Kingdom Brain Bank.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Age at disease onset | At enrolment
  Patients age when the initial symptom appeared.
Time to diagnosis | At enrolment
  Duration, in years, from appearance of initial symptom to receiving Parkinson's disease diagnosis.
Initial motor symptom | At enrolment
  Number of patients with each initial motor symptom (tremor, rigidity, or bradykinesia).
Side of initial motor symptoms | At enrolment
  Number of patients with either right or left side initial motor symptoms.
Clinical subtype of the disease | At enrolment
  Number patients with each disease subtype (tremor dominant Parkinson's disease, hypokinetic-rigid dominant Parkinson's disease, or postural instability and gait disturbance dominant Parkinson's disease).
Duration of levodopa treatment from disease onset | At enrolment
  Number of years on levodopa treatment since receiving parkinson's disease diagnosis
Levodopa equivalent dose | At enrolment
  Current dose of levodopa per day
Non-motor symptoms | At enrolment
  Non-motor symptoms measured by the non-motor symptoms questionnaire (NMS)
Quality of life | At enrolment
  Mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort assessed by the parkinson's disease quality of life questionnaire (PDQ-39).

SECONDARY OUTCOMES:
Stage of the disease [optional] | At enrolment
  The stage of the disease (stage 1, stage 2, stage 3, or stage 4) according to Hoehn and Yahr classification.
Motor Functions [optional] | At enrolment
  Motor functions assessed by the third part of the unified parkinson's disease rating scale (UPDRS III).

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be collected on a secure database (REDCap of Al-Azhar University). Investigators, who want to share a part of the whole of the patient data, should submit a request to our website (http://emra-collaborative.org/contact.html). They will enter in a data sharing agreement with the Egyptian National Research Collaborative to ensure proper acknowledgement of all study collaborators as non-author contributors in secondary publications from these data.

REFERENCES:
- [Background] Obeso JA, Rodriguez-Oroz MC, Benitez-Temino B, Blesa FJ, Guridi J, Marin C, Rodriguez M. Functional organization of the basal ganglia: therapeutic implications for Parkinson's disease. Mov Disord. 2008;23 Suppl 3:S548-59. doi: 10.1002/mds.22062. PMID 18781672
- [Background] Ceravolo R, Frosini D, Rossi C, Bonuccelli U. Impulse control disorders in Parkinson's disease: definition, epidemiology, risk factors, neurobiology and management. Parkinsonism Relat Disord. 2009 Dec;15 Suppl 4:S111-5. doi: 10.1016/S1353-8020(09)70847-8. PMID 20123548
- [Background] Blin P, Dureau-Pournin C, Foubert-Samier A, Grolleau A, Corbillon E, Jove J, Lassalle R, Robinson P, Poutignat N, Droz-Perroteau C, Moore N. Parkinson's disease incidence and prevalence assessment in France using the national healthcare insurance database. Eur J Neurol. 2015 Mar;22(3):464-71. doi: 10.1111/ene.12592. Epub 2014 Nov 12. PMID 25389031
- [Background] Durmus H, Gokalp MA, Hanagasi HA. Prevalence of Parkinson's disease in Baskale, Turkey: a population based study. Neurol Sci. 2015 Mar;36(3):411-3. doi: 10.1007/s10072-014-1988-x. Epub 2014 Oct 29. PMID 25351343
- [Background] Van Den Eeden SK, Tanner CM, Bernstein AL, Fross RD, Leimpeter A, Bloch DA, Nelson LM. Incidence of Parkinson's disease: variation by age, gender, and race/ethnicity. Am J Epidemiol. 2003 Jun 1;157(11):1015-22. doi: 10.1093/aje/kwg068. PMID 12777365
- [Background] Goetz CG, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stebbins GT, Stern MB, Tilley BC, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, Van Hilten JJ, LaPelle N. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Process, format, and clinimetric testing plan. Mov Disord. 2007 Jan;22(1):41-7. doi: 10.1002/mds.21198. PMID 17115387
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Liu WM, Wu RM, Lin JW, Liu YC, Chang CH, Lin CH. Time trends in the prevalence and incidence of Parkinson's disease in Taiwan: A nationwide, population-based study. J Formos Med Assoc. 2016 Jul;115(7):531-8. doi: 10.1016/j.jfma.2015.05.014. Epub 2015 Jun 27. PMID 26123636
- [Background] Pringsheim T, Jette N, Frolkis A, Steeves TD. The prevalence of Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2014 Nov;29(13):1583-90. doi: 10.1002/mds.25945. Epub 2014 Jun 28. PMID 24976103
- [Background] Douglas MR. Gene therapy for Parkinson's disease: state-of-the-art treatments for neurodegenerative disease. Expert Rev Neurother. 2013 Jun;13(6):695-705. doi: 10.1586/ern.13.58. PMID 23739006
- [Background] Wang G, Li XJ, Hu YS, Cheng Q, Wang CF, Xiao Q, Liu J, Ma JF, Zhou HY, Pan J, Tan YY, Wang Y, Chen SD. Mortality from Parkinson's disease in China: Findings from a five-year follow up study in Shanghai. Can J Neurol Sci. 2015 Jul;42(4):242-7. doi: 10.1017/cjn.2015.49. PMID 26153040
- [Background] Wright Willis A, Evanoff BA, Lian M, Criswell SR, Racette BA. Geographic and ethnic variation in Parkinson disease: a population-based study of US Medicare beneficiaries. Neuroepidemiology. 2010;34(3):143-51. doi: 10.1159/000275491. Epub 2010 Jan 15. PMID 20090375
- [Derived] Shaheen M, Mokarrab M, Youssef A, Aref M, Abushouk AI, Elmaraezy A, Almasswary A. Physiological evaluation of the provisional side-branch intervention strategy for bifurcation lesions using instantaneous wave-free ratio. Indian Heart J. 2018 Dec;70 Suppl 3(Suppl 3):S254-S258. doi: 10.1016/j.ihj.2018.01.028. Epub 2018 Jan 31. PMID 30595269